CLINICAL TRIAL: NCT03460353
Title: Bariatric Surgery and Pharmacokinetics Dexamphetamine: BAR-MEDS Dexamphetamine
Brief Title: Bariatric Surgery and Pharmacokinetics of Dexamphetamine
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Volvat Medisinsk Senter Stokkan (Other); Namsos Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1145i
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Morbid
Keywords: Bariatric surgery; Gastrointestinal tract; Biological availability; Pharmacokinetics; Dextroamphetamine
MeSH Terms: conditions — Obesity, Morbid | interventions — Dextroamphetamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dexamphetamine — Patients are tested for their normal prescription dexamphetamine medication
  Other Names: Dextroamphetamine

SUMMARY:
Changes to gastric pH, gastric emptying time, gastrointestinal transit-time or the pre-systemic metabolizing effect of enzymes secreted in the mucosa may all alter the pharmacokinetics of medicines. These factors are potentially influenced by bariatric surgery. Little is so far known about how gastric bypass and sleeve gastrectomy impacts the biological availability of medication. In this study the pharmacokinetic effects of bariatric surgery on dexamphetamine are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Preparing to undergo gastric bypass or sleeve gastrectomy in Central Norway
* Being a Norwegian citizen

Exclusion Criteria:

* Having previously undergone resections in the GI-tract

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for bariatric surgery (gastric bypass or sleeve gastrectomy)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Dexamphetamine concentration in blood serum (area under curve (AUC)) | From baseline to 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Strømmen, MSc, Principal Investigator — St. Olavs University Hospital
Locations (1):
- St. Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03460353/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03460353/SAP_001.pdf